CLINICAL TRIAL: NCT05388708
Title: ARDS in Children and ECMO Initiation Strategies Impact on Neurodevelopment (ASCEND)
Acronym: ASCEND
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ryan Barbaro, Associate Professor of Pediatrics, University of Michigan
Other Study IDs: HUM00173031; R01HL153519-01 (NIH)
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome; Extracorporeal Membrane Oxygenation
Keywords: ARDS; Acute Respiratory Distress Syndrome; Extracorporeal Membrane Oxygenation; ECMO; Extracorporeal Life Support; ECLS; Pediatric; Quality of Life; Functional Status
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual care ECMO Cohort: The cohort will be comprised of 550 patients, aged 14 days to 20 years, who go on extracorporeal membrane oxygenation (ECMO) support due to pediatric acute respiratory distress syndrome (PARDS) at physician discretion. Patients with qualifying PARDS must have one oxygenation index (OI) ≥ 16 or two OIs 12 ≥ to < 16 (at least 4 hours apart) or two oxygenation saturation indexes (OSIs) ≥ 10 (at least 4 hours apart) or one OI 12 ≥ to < 16 and one OSI > 10 (at least 4 hours apart) Subjects must be on mechanical ventilation for less than 240 hours (10 days) prior to cannulation. These measures must be after endotracheal intubation and before ECMO start. Chest radiograph prior to ECMO must show bilateral lung disease.
  Subjects cannulated on ECMO for no more than 96 hours prior to gaining consent.
  Interventions: Device: ECMO support
- PROSpect protocolized therapies cohort: The cohort will be comprised of 1000 patients, aged 14 days to 20 years, who are endotracheally intubated for PARDS. Patients with qualifying PARDS must have one oxygenation index (OI) ≥ 16 or two OIs 12 ≥ to < 16 (at least 4 hours apart) or two oxygenation saturation indexes (OSIs) ≥ 10 (at least 4 hours apart) or one OI 12 ≥ to < 16 and one OSI > 10 (at least 4 hours apart). These measures must be after endotracheal intubation. Chest radiograph must show bilateral lung disease. Patient must be enrolled in a clinical trial Prone and Oscillation Pediatric Clinical Trial (PROSpect) NCT01515787 which is distinct from ASCEND.
  PROSpect is a response adaptive randomized clinical trial, testing the impact of supine/prone positioning and conventional mechanical ventilation/high-frequency oscillatory ventilation on short and long-term clinical outcomes in children with severe PARDS. PROSpect manages severe PARDS subjects using a rigorous protocol that reserves ECMO for protocol failure.
  Interventions: Other: PROSpect protocolized therapies

INTERVENTIONS:
Device: ECMO support — ECMO prescribed by treating physicians for respiratory support in the setting of PARDS.
  Groups: Usual care ECMO Cohort
Other: PROSpect protocolized therapies — PROSpect is testing the impact of supine/prone positioning and conventional mechanical ventilation (CMV)/high-frequency oscillatory ventilation (HFOV) on clinical outcomes in 1,000 children with severe PARDS. PROSpect manages severe PARDS subjects using a protocol that reserves ECMO for protocol failure.
  The CMV group targets an exhaled tidal volume of 5-7mL/kg of ideal body weight and a peak inspiratory pressure <28 cm of H2O. The positive end expiratory pressure (PEEP) and FiO2 are titrated by a PEEP-FiO2 titration grid. The HFOV group titrates the mean airway pressure to target a FiO2 < 0.5 and a goal hemoglobin oxygen saturation of 88-92%. The frequency is titrated between 8-12 Hz and amplitude from 60-90 to achieve a goal pH of 7.15-7.30. Ventilation protocols are implemented until 28 days or extubation. Children randomized to the prone positioning will remain prone for at least 16 consecutive hours per day. Children randomized to supine positioning group remain supine.
  Groups: PROSpect protocolized therapies cohort

SUMMARY:
ASCEND researchers are partnering with families of children who receive extracorporeal membrane oxygenation (ECMO) after a sudden failure of breathing named pediatric acute respiratory distress syndrome (PARDS). ECMO is a life support technology that uses an artificial lung outside of the body to do the lung's work. ASCEND has two objectives.

The first objective is to learn more about children's abilities and quality of life among ECMO-supported children in the year after they leave the pediatric intensive care unit. The second objective is to compare short and long-term patient outcomes in two groups of children: one group managed with a mechanical ventilation protocol that reserves the use of extracorporeal membrane oxygenation (ECMO) until protocol failure to another group supported on ECMO per usual care.

DETAILED DESCRIPTION:
Decades after extracorporeal membrane oxygenation (ECMO) was first used to support children with severe pediatric acute respiratory distress syndrome (PARDS), pediatric intensivists lack both prospective studies of long-term outcomes in ECMO for PARDS and well-powered studies comparing the impact of ECMO initiation strategies on mortality and morbidity. While clinicians lack the equipoise necessary to randomize ECMO in dying children, there is uncertainty on if and when it is best to initiate ECMO to preserve survival, functioning, and quality of life. To determine if and when ECMO should be initiated in children with severe PARDS, it is necessary to compare the long-term outcomes in ECMO supported children to otherwise similar children who did not receive ECMO at the same threshold if at all.

An opportunity to address this question is provided by NHLBI-funded Prone and Oscillation Pediatric Clinical Trial (PROSpect) and the ECMO registry, Extracorporeal Life Support Organization (ELSO). PROSpect is an existing randomized clinical trial testing the impact of supine/prone positioning and conventional mechanical ventilation/high-frequency oscillatory ventilation on short and long-term clinical outcomes in 1,000 children with severe PARDS. PROSpect manages subjects with a rigorous protocol that reserves ECMO for protocol failure. The ELSO Registry includes children receiving usual care ECMO, initiated at the discretion of the intensivist.

ASCEND harmonizes PROSpect and ELSO data collection and prospectively measures functional status and quality of life via surveys in an additional 550 children with severe PARDS from ELSO sites. ASCEND measures children's abilities and quality of life when the child was in their normal state of health (just prior to being hospitalized), at discharge from the pediatric intensive care unit, and at 1-month, 3-months, 6-months, and 12-months after discharge from the pediatric intensive care unit. After enrollment of the usual care ECMO (in ELSO) and PROSpect's protocolized therapies (from the PROSpect clinical trial) is complete, then ASCEND will match similarly critically ill children based on their propensity to receive usual care ECMO.

ASCEND combines real-world observational data (from ELSO) and a randomized clinical trial (from PROSpect) to address two specific aims.

Aim 1: The study will test the hypotheses that one year after children receive usual care ECMO for PARDS, there will be a decline in long-term functional status and health-related quality of life as well as an increase in the proportion of children receiving respiratory support.

Aim 2: The study will test the hypotheses that 90-day mortality, one-year functional status, and one-year health-related quality of life are not equivalent for children with usual care ECMO (in ELSO) and PROSpect's protocolized therapies.

Protocol change in November 2021:

Inclusion criteria: Extend the window between intubation and ECMO cannulation from 120 hours to 168 hours.

Exclusion criteria: Remove active air leak, critical airway, and facial surgery/trauma within the last 2 weeks.

Protocol change in October 2022:

Inclusion criteria:

1. Extended the age range from 14 days - 17 years to 14 days - 20 years of age.
2. Extended the window between intubation and ECMO cannulation from 168 hours to 240 hours.

ELIGIBILITY:
Inclusion Criteria:

* Time between intubation and ECMO cannulation is less than 240 hours (10 days)
* ECMO support type is respiratory (VV or VA cannulation)
* Chest radiograph with bilateral lung disease
* Moderate or severe pediatric ARDS as measured by oxygenation index or oxygen saturation index after intubation and prior to ECMO cannulation:

One OI ≥ 16 or Two OIs ≥ 12 and ≤ 16 at least four hours apart or Two OSIs ≥ 10 at least four hours apart or One OI ≥ 12 and ≤ 16 and One OSI ≥ 10 at least four hours apart

Exclusion Criteria:

* Previously enrolled in PROSpect
* Perinatal related lung disease
* Congenital diaphragmatic hernia or congenital/acquired diaphragm paralysis
* Respiratory failure caused by cardiac failure or fluid overload
* Cyanotic congenital heart disease
* Cardiomyopathy
* Primary pulmonary hypertension (PAH)
* Unilateral lung disease
* Intubated for status asthmaticus
* Obstructive airway disease
* Bronchiolitis obliterans
* Post hematopoietic stem cell transplant
* Post lung transplant
* Home ventilator dependent
* Neuromuscular respiratory failure
* Head trauma: (managed with hyperventilation)
* Intracranial bleeding
* Unstable spine, femur or pelvic fractures
* Acute abdominal process/open abdomen
* Family/medical team have decided to not provide full support
* Enrolled in interventional clinical trial: not approved for co-enrollment; does not include cancer protocols.
* Known pregnancy

Ages: 14 Days to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population comes from pediatric patients hospitalized for respiratory distress requiring intubation and ECMO. Namely, children are eligible if they have moderate to severe PARDS, meet inclusion criteria and do not have the exclusion criteria listed below under exclusion criteria. Children in ELSO's usual care ECMO cohort also cannot be enrolled in PROSpect, and they must have respiratory ECMO initiated at an ELSO site within 10 days of intubation.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in functional status | baseline and 1 year after pediatric intensive care unit discharge
  This primary natural history outcome is measured among usual care extracorporeal membrane oxygenation (ECMO) patients. This outcome is the change in functional status as measured at baseline and 12 months after pediatric intensive care unit (PICU) discharge. The instrument is the functional status scale score. The baseline measure will be made within 96 hours of ECMO initiation and reflect patient's status in the week prior to ECMO.
  The Functional Status Scale (FSS) is a valid and reliable assessment method to quantify functional status. The FSS includes 6 domains: mental status, sensory functioning, communication, motor function, feeding, and respiratory. Scores for each domain range from 1 (normal) to 5 (very severe dysfunction); total scores range from 6 to 30 with higher scores reflecting worse functioning.
Change in health-related quality of life | baseline and 1 year after pediatric intensive care unit discharge
  This primary natural history outcome is measured among usual care ECMO patients. This outcome is the change in the health-related quality of life as measured at baseline and 12 months after PICU discharge. The instrument is the age-appropriate Version 4.0 Pediatric Quality of Life Inventory (PedsQL 4.0) generic core scales for acute illness.
  PedsQL 4.0 Generic Core Scales and Infant Scales - Acute Version are parent proxy-report scales. The scales ranges from 0 to 100, with higher scores indicating fewer problems. PedsQL 4.0 Generic Core Scales is a 23-item scale with 4 domains: physical functioning, emotional functioning, social functioning, and school functioning. The PedsQL Infant Scales consist of 36-45 questions, depending on age, with 5 domains: physical functioning, physical symptoms, emotional functioning, social functioning, and cognitive functioning.
The proportion of children with a new morbidity | baseline and 1 year after pediatric intensive care unit discharge
  This primary natural history outcome is measured among usual care ECMO patients. A new morbidity is defined as a change in the functional status scale score instrument by 3 or more, as previously described. This outcome will report the proportion of children who acquire a new morbidity as measured at baseline and 12 months after PICU discharge.
  The Functional Status Scale (FSS) is a valid and reliable assessment method to quantify functional status. The FSS includes 6 domains: mental status, sensory functioning, communication, motor function, feeding, and respiratory. Scores for each domain range from 1 (normal) to 5 (very severe dysfunction); total scores range from 6 to 30 with higher scores reflecting worse functioning.
All-cause mortality at hospital discharge or 90-days | 90 days after the day of illness on which patients from the two cohorts are matched
  This primary comparative short-term outcome is measured among both usual care ECMO and Prone and Oscillation Pediatric Clinical Trial (PROSpect) protocolized therapy groups. The outcome compares the 90-day mortality for matched children in the two groups. The endpoint is 90 days after the day of illness on which patients from the two cohorts are matched or hospital discharge.
Comparative change in one-year functional status | baseline and 1 year after pediatric intensive care unit discharge
  This primary comparative long-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. The outcome compares the change in the functional status as measured at baseline and 12 months after PICU discharge between matched children in the two groups. The instrument is the functional status scale score.
  The Functional Status Scale (FSS) is a valid and reliable assessment method to quantify functional status. The FSS includes 6 domains: mental status, sensory functioning, communication, motor function, feeding, and respiratory. Scores for each domain range from 1 (normal) to 5 (very severe dysfunction); total scores range from 6 to 30 with higher scores reflecting worse functioning.
Comparative change in one-year health-related quality of life | baseline and 1 year after pediatric intensive care unit discharge
  This primary comparative long-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. The outcome compares the change in the health-related quality of life as measured at baseline and 12 months after PICU discharge between matched children in the two groups. The instrument is the change in the age-appropriate PedsQL 4.0 generic core scales for acute illness.
  PedsQL 4.0 Generic Core Scales and Infant Scales - Acute Version are parent proxy-report scales. The scales ranges from 0 to 100, with higher scores indicating fewer problems. PedsQL 4.0 Generic Core Scales is a 23-item scale with 4 domains: physical functioning, emotional functioning, social functioning, and school functioning. The PedsQL Infant Scales consist of 36-45 questions, depending on age, with 5 domains: physical functioning, physical symptoms, emotional functioning, social functioning, and cognitive functioning.

SECONDARY OUTCOMES:
Change in pediatric overall performance category | baseline and 1 year after pediatric intensive care unit discharge
  This secondary natural history outcome is measured among usual care ECMO patients. The outcome is the change in the pediatric overall performance category measured at baseline and 12 months after PICU discharge. The instrument is the pediatric overall performance category.
  The Pediatric Overall Performance Category (POPC) quantifies impairments and functional morbidity. Scores range from 1 to 6 with 1: good, 2: mild disability, 3: moderate disability, 4: severe disability, 5: coma, and 6: brain death.
Change in pediatric cerebral performance category | baseline and 1 year after pediatric intensive care unit discharge
  This secondary natural history outcome is measured among usual care ECMO patients. This outcome is the change in the pediatric cerebral performance category measured at baseline and 12 months after PICU discharge. The instrument is the pediatric cerebral performance category.
  The Pediatric Cerebral Performance Category (PCPC) quantifies cognitive impairments. Scores range from 1 to 6 with 1: good, 2: mild disability, 3: moderate disability, 4: severe disability, 5: coma, and 6: brain death.
Change in breathing support | baseline and 1 year after pediatric intensive care unit discharge
  This secondary natural history outcome is measured among usual care ECMO patients. This outcome is the change in breathing support measured at baseline and 12 months after PICU discharge. The instrument is the respiratory subscale of the functional status scale score.
  The Functional Status Scale (FSS) is a valid and reliable assessment method to quantify functional status with 6 domains. This measure of breathing support will rely on the FSS respiratory domain. The respiratory domain score ranges from 1 (normal) to 5 (very severe dysfunction).
Change in the psychosocial component of health-related quality of life | baseline and 1 year after pediatric intensive care unit discharge
  This secondary natural history outcome is measured among usual care ECMO patients. This outcome is the change in the psychosocial component of health-related quality of life measured at baseline and 12 months after PICU discharge. The instrument is the age-appropriate psychosocial health summary score of the PedsQL 4.0 generic core scales for acute illness.
  PedsQL 4.0 Generic Core Scales and Infant Scales - Acute Version are parent proxy-report scales. The scales range from 0 to 100, with higher scores indicating fewer problems. The psychosocial component of the PedsQL 4.0 Generic Core Scales is composed of three of the four domains: emotional functioning, social functioning, and school functioning. The PedsQL Infant Scales psychosocial component is composed of three of the five domains: emotional functioning, social functioning, and cognitive functioning.
Change in the physical component of health-related quality of life | baseline and 1 year after pediatric intensive care unit discharge
  This secondary natural history outcome is measured among usual care ECMO patients. The outcome is the change in the physical component of health-related quality of life measured at baseline and 12 months after PICU discharge. The instrument is the age-appropriate physical health summary score of the PedsQL 4.0 generic core scales for acute illness.
  PedsQL 4.0 Generic Core Scales and Infant Scales - Acute Version are parent proxy-report scales. The scales range from 0 to 100, with higher scores indicating fewer problems. The physical component of the PedsQL 4.0 Generic Core Scales is composed of one of the four domains: physical functioning. The PedsQL Infant Scales physical component is composed of two of the five domains: physical functioning and physical symptoms.
Change in child fatigue | baseline and 1 year after pediatric intensive care unit discharge
  This secondary natural history outcome is measured among usual care ECMO patients. This outcome is the change in child fatigue measured at baseline and 12 months after PICU discharge. The instrument is the age-appropriate PedsQL fatigue scale for acute illness.
  The PedsQL™ Multi-dimensional Fatigue Scale - Acute Version is an 18-item scale that encompasses three domains: General Fatigue, Sleep/Rest Fatigue and Cognitive Fatigue. The scale ranges from 0 to 100, with higher scores indicating fewer problems and better health-related quality of life.
Change in family impact of the child's health | baseline and 1 year after pediatric intensive care unit discharge
  This secondary natural history outcome is measured among usual care ECMO patients. This outcome is the change in child fatigue measured at baseline and 12 months after PICU discharge. The instrument is the age-appropriate PedsQL fatigue scale for acute illness.
  The PedsQL™ Family Impact Module - Acute Version is a 36-item scale that encompasses eight domains: Physical Functioning, Emotional Functioning, Social Functioning, Cognitive Functioning, Communication, Worry, Daily Activities, and Family Relationships. The scale ranges from 0 to 100, with higher scores indicating fewer problems.
Change in one-year functional status of children suffering a neurologic injury | baseline and 1 year after pediatric intensive care unit discharge
  This secondary natural history outcome is measured among usual care ECMO patients. A neurologic injury is defined as a new intracranial hemorrhage or stroke recognized on radiologic imaging. This outcome will compare the change in functional status as measured at baseline and 12 months after PICU discharge between those children who suffered a neurologic injury to those who did not. The instrument is the functional status scale score.
  The Functional Status Scale (FSS) is a valid and reliable assessment method to quantify functional status. The FSS includes 6 domains: mental status, sensory functioning, communication, motor function, feeding, and respiratory. Scores for each domain range from 1 (normal) to 5 (very severe dysfunction) with total scores ranging from 6 to 30.
Difference between groups in intracranial bleeding or ischemic stroke | 28 days after day in illness patients are matched or during hospitalization
  This secondary comparative short-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. This outcome compares the difference in the proportion of matched children who suffer a new intracranial hemorrhage or ischemic stroke (recognized on radiologic imaging) between the two groups.
Difference between groups in pneumothorax | 28 days after day in illness patients are matched or during hospitalization
  This secondary comparative short-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. This outcome compares the difference in the proportion of matched children who suffer a pulmonary complication of a new pneumothorax at 28 days between children in the two groups.
Comparative difference in the change in child fatigue | baseline and 1 year after pediatric intensive care unit discharge
  This secondary comparative long-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. This outcome compares the change in child fatigue as measured at baseline and 12 months after PICU discharge between matched children in the two groups. The instrument is the age-appropriate PedsQL fatigue scale for acute illness.
  The PedsQL™ Multi-dimensional Fatigue Scale - Acute Version is an 18-item scale that encompasses three domains: General Fatigue, Sleep/Rest Fatigue and Cognitive Fatigue. The scale ranges from 0 to 100, with higher scores indicating fewer problems and better health-related quality of life.
Comparative difference in the change in family impact of the child's health | baseline and 1 year after pediatric intensive care unit discharge
  This secondary comparative long-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. This outcome compares the change in family impact of the child's health as measured at baseline and 12 months after PICU discharge between matched children in the two groups. The instrument is the PedsQL family impact module for acute illness.
  The PedsQL™ Family Impact Module - Acute Version is a 36-item scale that encompasses eight domains: Physical Functioning, Emotional Functioning, Social Functioning, Cognitive Functioning, Communication, Worry, Daily Activities, and Family Relationships. The scale ranges from 0 to 100, with higher scores indicating fewer problems.
Comparative difference in the change in the psychosocial component of health-related quality of life | baseline and 1 year after pediatric intensive care unit discharge
  This secondary comparative long-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. This outcome compares the change in the psychosocial component of health-related quality of life as measured at baseline and 12 months after PICU discharge between matched children in the two groups. The instrument is the age-appropriate psychosocial health summary score from PedsQL 4.0 generic core scales for acute illness.
  PedsQL 4.0 Generic Core Scales and Infant Scales - Acute Version are parent proxy-report scales. The scale ranges from 0 to 100, with higher scores indicating fewer problems. The psychosocial component of the PedsQL 4.0 Generic Core Scales is composed of three of the four domains: emotional functioning, social functioning, and school functioning. The PedsQL Infant Scales psychosocial component is composed of three of the five domains: emotional functioning, social functioning, and cognitive functioning.
Comparative difference in the in change in the physical component of health-related quality of life | baseline and 1 year after pediatric intensive care unit discharge
  This secondary comparative long-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. This outcome compares the change in the physical component of health-related quality of life as measured at baseline and 12 months after PICU discharge between matched children in the two groups. The instrument is the age-appropriate physical health summary score from PedsQL 4.0 generic core scales for acute illness.
  PedsQL 4.0 Generic Core Scales and Infant Scales - Acute Version are parent proxy-report scales. The scales range from 0 to 100, with higher scores indicating fewer problems. The physical component of the PedsQL 4.0 Generic Core Scales is composed of one of the four domains: physical functioning. The PedsQL Infant Scales physical component is composed of two of the five domains: physical functioning and physical symptoms.
Comparative change in respiratory support | baseline and 1 year after pediatric intensive care unit discharge
  This secondary comparative long-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. This outcome compares the change in respiratory support as measured at baseline and 12 months after PICU discharge between matched children in the two groups. The instrument is the respiratory subscale of the functional status scale score.
  The Functional Status Scale (FSS) is a valid and reliable assessment method to quantify functional status with 6 domains. This measure of breathing support will rely on the FSS respiratory domain. The respiratory domain score ranges from 1 (normal) to 5 (very severe dysfunction).
Comparative difference in new morbidity | baseline and 1 year after pediatric intensive care unit discharge
  This secondary comparative long-term outcome is measured among both usual care ECMO and PROSpect protocolized therapy groups. A new morbidity is defined as a change in the functional status scale instrument score by 3 or more, as previously described. This outcome compares the change in the proportion of matched children who acquire a new morbidity as measured at baseline and 12 months after PICU discharge between the two groups.
  The Functional Status Scale is a valid and reliable assessment method to quantify functional status. The FSS includes 6 domains: mental status, sensory functioning, communication, motor function, feeding, and respiratory. Scores for each domain range from 1 (normal) to 5 (very severe dysfunction) with total scores ranging from 6 to 30.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Barbaro, MD, Principal Investigator — University of Michigan
Locations (99):
- United States (76):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Children's Hospital, Loma Linda, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - UCSF Benioff Children's Hospital - San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Nemours Children's Hospital, Delaware, Wilmington, Delaware
  - UF Health Shands Children's Hospital, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Orlando Health Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Florida, Orlando, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Kapi'olani Medical Center for Women & Children, Honolulu, Hawaii
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Comer Children's Hospital, Chicago, Illinois
  - OSF Healthcare Children's Hospital of Illinois, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Health Care Stead Family Children's Hospital, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner LSU Health Shreveport, Shreveport, Louisiana
  - University of Maryland Children's Hospital, Baltimore, Maryland
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Minnesota Hospital, Minneapolis, Minnesota
  - M Health Fairview Masonic Children's Hospital, Minneapolis, Minnesota
  - Mayo Eugenio Litta Children's Hospital, Rochester, Minnesota
  - Children's Mercy, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Nebraska, Omaha, Nebraska
  - UNM Children's Hospital, Albuquerque, New Mexico
  - John R. Oishei Children's Hospital, Buffalo, New York
  - Hassenfeld Children's Hospital at NYU Langone, New York, New York
  - NewYork-Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - NewYork-Presbyterian Komansky Children's Hospital, New York, New York
  - Cohen Children's Medical Center, Queens, New York
  - N.C. Children's Hospital, Chapel Hill, North Carolina
  - Duke Children's Hospital & Health Center, Durham, North Carolina
  - Atrium Health Wake Forest Baptist | Brenner Children's Hospital, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma Children's Hospital OU Health, Oklahoma City, Oklahoma
  - OHSU Doernbecher Children's Hospital, Portland, Oregon
  - Penn State Health Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hasbro Children's, Providence, Rhode Island
  - MUSC Shawn Jenkins Children's Hospital, Charleston, South Carolina
  - Sanford Children's Hospital, Sious Falls, South Dakota
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Dell Children's Medical Center, Austin, Texas
  - Medical City Children's Hospital, Dallas, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Children's Memorial Hermann Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - University Health Women's & Children's Hospital, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - UVA Children's Hospital, Charlottesville, Virginia
  - Inova L.J. Murphy Children's Hospital, Falls Church, Virginia
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - UW Health American Family Children's Hospital, Madison, Wisconsin
  - Children's Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - The Royal Children's Hospital Melbourne, Melbourne
  - Perth Children's Hospital, Perth
  - Queensland Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario
- Pontificia Universidad, Santiago, Chile
- Fundacion Cardiovascular De Colombia, Floridablanca, Colombia
- Istituto Giannina Gaslini, Genoa, Italy
- Starship Children's Hospital, Grafton, Aukland, New Zealand
- Hospital de Santa Maria, Lisbon, Portugal
- Spain (3):
  - Children's Hospital and Vall d' Hebron Women's Hospital, Barcelona
  - Sant Joan de Deu Barcelona Hospital, Barcelona
  - Hospital Gregorio Maranon, Madrid
- ECMO Centrum Karolinska, Stockholm, Sweden
- United Kingdom (8):
  - Royal Hospital for Children, Glasgow
  - Leicester Children's Hospital, Leicester
  - Alder Hey Children's Hospital, Liverpool
  - Evelina London Children's Hospital, London
  - Royal Brompton Hospital, London
  - Great Ormond Street Hospital for Children, London
  - Freeman Hospital, Newcastle upon Tyne
  - Southampton Children's Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
It is the National Institutes of Health (NIH) policy that the results and accomplishments of the activities that it funds should be made available to the public (see https://grants.nih.gov/policy/sharing.htm).
  After the study is completed, the de-identified, archived data will be transmitted to and stored at the Biologic Specimen and Data Repository Information Coordination Center (BioLINCC), for use by other researchers including those outside of the study. Permission to transmit data to the BioLINCC will be included in the informed consent.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Two years after study analysis is complete.
Access Criteria: ASCEND investigators will compose the ASCEND steering committee lead by PI Barbaro. Members include Ryan Barbaro, Theodore Iwashyna, Martha Curley, Carol Hodgson, Seth Warschausky and Ben Hansen. The steering committee will be responsible for developing publication procedures and resolving authorship issues.

REFERENCES:
- [Background] Fiser DH. Assessing the outcome of pediatric intensive care. J Pediatr. 1992 Jul;121(1):68-74. doi: 10.1016/s0022-3476(05)82544-2. PMID 1625096
- [Background] Pollack MM, Holubkov R, Glass P, Dean JM, Meert KL, Zimmerman J, Anand KJ, Carcillo J, Newth CJ, Harrison R, Willson DF, Nicholson C; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Functional Status Scale: new pediatric outcome measure. Pediatrics. 2009 Jul;124(1):e18-28. doi: 10.1542/peds.2008-1987. PMID 19564265
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] Pollack MM, Holubkov R, Funai T, Berger JT, Clark AE, Meert K, Berg RA, Carcillo J, Wessel DL, Moler F, Dalton H, Newth CJ, Shanley T, Harrison RE, Doctor A, Jenkins TL, Tamburro R, Dean JM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network. Simultaneous Prediction of New Morbidity, Mortality, and Survival Without New Morbidity From Pediatric Intensive Care: A New Paradigm for Outcomes Assessment. Crit Care Med. 2015 Aug;43(8):1699-709. doi: 10.1097/CCM.0000000000001081. PMID 25985385
- [Background] Keim G, Watson RS, Thomas NJ, Yehya N. New Morbidity and Discharge Disposition of Pediatric Acute Respiratory Distress Syndrome Survivors. Crit Care Med. 2018 Nov;46(11):1731-1738. doi: 10.1097/CCM.0000000000003341. PMID 30024428
- [Background] Combes A, Hajage D, Capellier G, Demoule A, Lavoue S, Guervilly C, Da Silva D, Zafrani L, Tirot P, Veber B, Maury E, Levy B, Cohen Y, Richard C, Kalfon P, Bouadma L, Mehdaoui H, Beduneau G, Lebreton G, Brochard L, Ferguson ND, Fan E, Slutsky AS, Brodie D, Mercat A; EOLIA Trial Group, REVA, and ECMONet. Extracorporeal Membrane Oxygenation for Severe Acute Respiratory Distress Syndrome. N Engl J Med. 2018 May 24;378(21):1965-1975. doi: 10.1056/NEJMoa1800385. PMID 29791822